CLINICAL TRIAL: NCT06799403
Title: Stop for Stress - En Sammenligning af Online og Gruppebaseret Behandling for Arbejdsrelateret Stress
Brief Title: Stop for Stress - a Randomized Controlled Trial Comparing an Online and a Group-based Format of an Intervention for Work-related Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lea Nørgaard Sørensen (Other)
Collaborators: Gødstrup Hospital (Other)
Responsible Party: Sponsor-Investigator, Lea Nørgaard Sørensen, PhD student, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-108-24
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Work-Related Stress
Keywords: work-related stress; online intervention; group intervention; return-to-work
MeSH Terms: conditions — Occupational Stress | interventions — Mars

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapist-assisted online delivery format (Experimental): Participants will gain access to an online program comprised by 14 modules covering psychoeducation on stress, sleep, and communication, cognitive behavioral restructuring, and exercises and tools for dealing with stress and preventing relapse. Participants are followed by a therapist providing feedback on exercises and progress. The program extends over approx. 12 weeks.
  Interventions: Behavioral: Therapist-assisted online stress management
- Group-based face-to-face delivery format (Active Comparator): The group-based format consists of 8 sessions of each 3 hours spread across 12 weeks. The sessions cover psychoeducation on stress, sleep, and communication, cognitive behavioral restructuring, and exercises and tools for dealing with stress and preventing relaps. A group includes 8-9 participants
  Interventions: Behavioral: Group-based face-to-face stress management

INTERVENTIONS:
Behavioral: Therapist-assisted online stress management — Participants gain access to an online program comprised by 14 modules covering psychoeducation on stress, sleep, and communication, cognitive behavioral restructuring, and exercises and tools for dealing with stress and preventing relapse. Participants are followed by a therapist providing feedback on exercises and progress. The program extends over approx. 12 weeks.
  Other Names: Stop for Stress
  Arms: Therapist-assisted online delivery format
Behavioral: Group-based face-to-face stress management — The group-based format consists of 8 sessions of each 3 hours spread across 12 weeks. The sessions cover psychoeducation on stress, sleep, and communication, cognitive behavioral restructuring, and exercises and tools for dealing with stress and preventing relaps. A group includes 8-9 participants
  Other Names: MARS
  Arms: Group-based face-to-face delivery format

SUMMARY:
Work-related stress is a major public health concern, causing sickness absenteeism and impaired health and well-being. Many afflicted with severe work-related stress will not receive evidence-based treatment due to geographical distance, stigma and unwillingness to participate in a group, creating unequality access to healthcare services. Online interventions show comparable effects to face-to-face interventions and have potential to break down some of these barriers. We have developed and pilot tested the online delivery format of the intervention for work-related stress, Stop for Stress, with promising results. In a two-armed, multicentre randomized controlled trial we aim to 1) compare the effect of the online delivery format and an evidence-based face-to-face group-based format and 2) identify markers of enhanced outcomes in each delivery format. The study will include 220 patients with severe work-related stress (110 from each of two centres) who are randomizes 1:1 to the two interventions. Outcomes consist of self-report measures of psychological symptoms, cognitive functioning, sleep, and perceived working environment and register data on ebsenteeism and return-to-work.

ELIGIBILITY:
Inclusion Criteria:

* Current employment and significant work-related stressors
* Perceived Stress Scale (PSS-10) score ≥20 and symptom duration >4 weeks
* In case of full-time sick leave, return to work must be planned concurrent with the intervention
* Access to a computer or tablet with internet connection at home

Exclusion Criteria:

* Interpersonal difficulties, bullying, harassment, violence, threats, and traumatic events as primary stressor
* Severe stressors outside of work
* Symptoms meeting diagnostic criteria for anxiety, depression or severe psychiatric illnesses requiring specialized treatment
* Current abuse of alcohol and/or psychoactive drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Perceived stress (T1) | Post intervention: 3 months from baseline
  Self-report measure using the 10 item Perceived Stress Scale (PSS-10), 10 items on a 0-4 scale, ranging from 0-40 point with higher scores indicating more perceived stress.
Obejctive cognitive functioning measures by ICAT (T2) | Follow-up: 6 months from baseline
  ICAT (Internet-Based Cognitive Assessment Tool) comprises 5 subtests (list learning, consonant repitition, letter-number sequencing, delayed list learning, visuomotor tracking)
Return-to-work | Participants are followed continously from 5 yeras prior to enrollment (baseline) and until 12 months follow-up
  Derived from the Danish national DREAM registry, comprising information on weekly transfer income (e.g. long-term sickness absence) and employment status

SECONDARY OUTCOMES:
Perceived Stress (T2) | Follow-up: 6 months from baseline
  Self-report measure using the 10 item Perceived Stress Scale (PSS-10), 10 items on a 0-4 scale, ranging from 0-40 point with higher scores indicating more perceived stress.
Perceived Stress (T3) | Follow-up: 12 months from baseline
  Self-report measure using the 10 item Perceived Stress Scale (PSS-10), 10 items on a 0-4 scale, ranging from 0-40 point with higher scores indicating more perceived stress.
Cognitive functioning (T1) | Post intervention: 3 months from baseline
  Self-report measure using the Cognitive Failures Questionnaire (CFQ), 25 items on a 0-4 point scale, range 0-100 with higher scores indicating lower subjective cognitive functioning.
Working environment (T1) | Post intervention: 3 months from baseline
  Perceived working environment self-reported using selected (independent) items from the Danish Psychosocial Questionnaire (DPQ). Includes influence, predictability, work load, relations to coworkers, relations to managers, recognition, and meaning.
Working environment (T2) | Follow-up: 6 months from baseline
  Perceived working environment self-reported using selected (independent) items from the Danish Psychosocial Questionnaire (DPQ). Includes influence, predictability, work load, relations to coworkers, relations to managers, recognition, and meaning.
Work ability (T1) | Post intervention: 3 months from baseline
  Self-report measure using the Work Ability Index (WAI), 1 item scale ranging from 0-10 with higher scores indicating better work ability
Work ability (T2) | Follow-up: 6 months from baseline
  Self-report measure using the Work Ability Index (WAI), 1 item scale ranging from 0-10 with higher scores indicating better work ability
Work ability (T3) | Follow-up: 12 months from baseline
  Self-report measure using the Work Ability Index (WAI), 1 item scale ranging from 0-10 with higher scores indicating better work ability

OTHER OUTCOMES:
Utilizations of psychotropic drug prescriptions | Participants are followed continously from 5 yeras prior to enrollment (baseline) and until 12 months follow-up
  Derived from the Danish national Register of Medical Products Statistics. Includes presciptions on antidepressants, anxiolytics, sedatives and anagesics.
Working environment (T3) | Follow-up: 12 months from baseline
  Perceived working environment self-reported using selected (independent) items from the Danish Psychosocial Questionnaire (DPQ). Includes influence, predictability, work load, relations to coworkers, relations to managers, recognition, and meaning.
Cognitive functioning (T2) | Follow-up: 6 months from baseline
  Self-reportmeasure using the Cognitive Failures Questionnaire (CFQ), 25 items on a 0-4 point scale, range 0-100 with higher scores indicating lower subjective cognitive functioning.
Symptoms of depression and anxiety (T1) | Post intervention: 3 months from baseline
  Self-report measure using the Common Mental Disorders Questionniare (CMDQ), 10 items in total: 4 item on the anxiety scale (0-4 point scale, range 0-16) and 6 items on the depression scale (0-4 point scale, range 0-24) with higher scores indicating more severe symptoms.
Symptoms of depression and axiety (T2) | Follow-up: 6 months from baseline
  Self-report measure using the Common Mental Disorders Questionniare (CMDQ), 10 items in total: 4 item on the anxiety scale (0-4 point scale, range 0-16) and 6 items on the depression scale (0-4 point scale, range 0-24) with higher scores indicating more severe symptoms.
Symptoms of depression and anxiety (T3) | Follow-up: 12 months from baseline
  Self-report measure using the Common Mental Disorders Questionniare (CMDQ), 10 items in total: 4 item on the anxiety scale (0-4 point scale, range 0-16) and 6 items on the depression scale (0-4 point scale, range 0-24) with higher scores indicating more severe symptoms.
Daily functioning (T3) | Follow-up: 12 months from baseline
  Self-report measure using the Work and Social Adjustment Scale (WSAS), 5 items 0-8 point scale, ranging from 0-40 point, where higher scores indicate more impaired daily functioning.
Daily functioning (T2) | Follow-up: 6 months from baseline
  Self-report measure using the Work and Social Adjustment Scale (WSAS), 5 items 0-8 point scale, ranging from 0-40 point, where higher scores indicate more impaired daily functioning.
Daily functioning (T1) | Post intervention: 3 months from baseline
  Self-report measure using the Work and Social Adjustment Scale (WSAS), 5 items 0-8 point scale, ranging from 0-40 point, where higher scores indicate more impaired daily functioning.
Cognitive functioning (T3) | Follow-up: 12 months from baseline
  Self-reportmeasure using the Cognitive Failures Questionnaire (CFQ), 25 items on a 0-4 point scale, range 0-100 with higher scores indicating lower subjective cognitive functioning.
Sleep quality (T1) | Post intervention: 3 months from baseline
  Self-report measure using the Basic Nordic Sleep Questionnaire (BSNQ), 7 items on a 1-5 scale, ranging from 7-35 points with higher scores indicating lower subjective sleep quality
Sleep quality (T2) | Follow-up: 6 months from baseline
  Self-report measure using the Basic Nordic Sleep Questionnaire (BSNQ), 7 items on a 1-5 scale, ranging from 7-35 points with higher scores indicating lower subjective sleep quality
Sleep quality (T3) | Follow-up: 12 months from baseline
  Self-report measure using the Basic Nordic Sleep Questionnaire (BSNQ), 7 items on a 1-5 scale, ranging from 7-35 points with higher scores indicating lower subjective sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Zara A Stokholm, MD, PhD, Principal Investigator — Department of Occupational and Environmental Medicine, Danish Ramazzini Centre, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Occupational and Environmental Medicine, Aarhus University Hospital, Aarhus, Central Region Denmark
  - Department of Occupational and Environmental Medicine, Gødstrup Hospital, Herning, Central Region Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willert MV, Thulstrup AM, Bonde JP. Effects of a stress management intervention on absenteeism and return to work--results from a randomized wait-list controlled trial. Scand J Work Environ Health. 2011 May;37(3):186-95. doi: 10.5271/sjweh.3130. Epub 2010 Nov 8. PMID 21057736
- See also: Danish project website that inform potentional participant and general practitioners about the aim of the study, who can participate, and what is expected of participants. — http://stopforstress.auh.dk